CLINICAL TRIAL: NCT02788565
Title: SOMATOSTATIN TREATMENT EXPERIENCE TRIAL An Observational Cross Sectional Trial Investigating Quality of Life, Treatment Experience and Direct Cost of Treatment With Somatostatin Analogues in Subjects With Gastroenteropancreatic Neuroendocrine Tumours (GEP-NETS)
Brief Title: Quality of Life, Treatment Experience and Cost of Treatment With Somatostatin Analogues in Patients With Gastroenteropancreatic Neuroendocrine Tumours
Acronym: STREET
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-SE-52030-353
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumours

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Data from this study will contribute additional knowledge regarding patient outcomes and direct somatostatin analogue (SSA) treatment related costs in clinical practice in the Nordic countries. Such knowledge can be of importance in a treatment decision, decision support for development of care, follow up and training of both patients and primary care nurses.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Diagnosed with a Gastroenteropancreatic Neuroendocrine Tumour (GEP-NET) and treated with SSA for at least three months but not more than 3 years
* GEP-NET proliferation index Ki 67 <10%
* Over 18 years of age

Exclusion Criteria:

* No specific exclusion criteria defined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment clinic
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with injection problems according to the subject | Day 1
  Subject questionnaire asks "In your opinion, how did the last injection go?", subject chooses either 'no problems' or 'problems occurred'.

SECONDARY OUTCOMES:
Quality of life, mean physical health score in SF-12 derived according to the SF-12 manual. | Day 1
  Mean physical health score and mean mental health score in SF-12 derived according to the SF-12 manual
Quality of life, mean mental health score in SF-12 derived according to the SF-12 manual. | Day 1
Subject experience: proportion of subjects reporting "much" or "very much" anxiety in subject questionnaire. | Day 1
  Subjects asked "To what extent do you feel anxiety before the injection?"
Mean number of packs of H01CB03 and H01CB02 purchased. | Retrospective data collection of a 1 year period
Median number of packs of H01CB03 and H01CB02 purchased. | Retrospective data collection of a 1 year period
Mean number of two consecutive dispensed prescriptions of H01CB03, H01CB02 within seven days during the pre-specified one-year period of retrospective data extraction. | Retrospective data collection of a 1 year period
Median number of two consecutive dispensed prescriptions of H01CB03, H01CB02 within seven days during the pre-specified one-year period of retrospective data extraction. | Retrospective data collection of a 1 year period
Median frequency of visits to treating physician in hospital will be derived as number of (frequency) of revisits recorded in the subject questionnaire. | Day 1
Median time - visits to primary care for injections; visits to treating physician at hospital; time to travel | Day 1
Median time for giving injections of SSA in subjects, derived as the time reported in the nurse questionnaire. | Day 1
Proportion of nurses who reported "moderately" or "very" or "very much" confidence in giving injections | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (2):
- Sweden (2):
  - Skane University Hospital, Lund
  - Uppsala University Hospital, Uppsala